CLINICAL TRIAL: NCT02481271
Title: Effects of Preoperative Relaxation and Intensified Surgery Education on Preoperative Wellbeing and Postoperative Complaints in Patients Undergoing Cholcystectomy - a Randomized Controlled Trial
Brief Title: Preoperative Relaxation and Intensified Patient Surgery Education in Patients Undergoing Cholecystectomy
Acronym: MBM_Galle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Gustav Dobos, Principle Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 14-6061-BO MBM_Galle
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Gall Stones
Keywords: cholecystectomy
MeSH Terms: conditions — Gallstones | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual care (No Intervention): Does not receive a specific study intervention
- preoperative relaxation program (Experimental): preoperative relaxation program
  Interventions: Behavioral: relaxation program
- preoperative surgery education (Experimental): single education unit to understand the complete surgical procedures
  Interventions: Behavioral: surgery education
- preoperative relaxation program+preoperative surgery education (Experimental): preoperative relaxation program AND single education unit
  Interventions: Behavioral: relaxation program; Behavioral: surgery education

INTERVENTIONS:
Behavioral: relaxation program — relaxation and mindfulness techniques such as body scan, breathing meditation or imagination exercises
  1 week program, one introductory session and daily home practice
  Arms: preoperative relaxation program; preoperative relaxation program+preoperative surgery education
Behavioral: surgery education — intensified education unit to reduce anxiety and stress, by using pictures and videos of rooms, and procedures of the planned surgery
  1 single unit in the week before the surgery
  Arms: preoperative relaxation program+preoperative surgery education; preoperative surgery education

SUMMARY:
This study aims to test the effects of a Preoperative Relaxation intervention and an Intensified Surgery Patient Education on pre- and postoperative wellbeing and health in Patients Undergoing Cholecystectomy.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* referral for cholecystectomy
* preoperative anxiety at least 4/10 points on a numeric rating scale
* physical and mental capability to participant
* written informed consent

Exclusion Criteria:

* Emergency surgery
* malignoma
* severe comorbidity
* severe psychological disorders
* immunosuppression
* coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | day of surgery
  State Anxiety (STAI-S) (Spielberger 1970)
postoperative pain intensity | day after the surgery, before meditation
  numeric rating scale for pain at rest, pain at mobilization, coughing, washing, breathing and moving

SECONDARY OUTCOMES:
preoperative anxiety | day of surgery
  Trait Anxiety (STAI-T) (Spielberger 1970)
preoperative anxiety | day of surgery
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) (Berth 2007)
preoperative anxiety | day of surgery
  Anaesthesia- and Surgery-dependent Preoperative Anxiety (ASPA) (Wetsch 2009)
postoperative disability | day after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative disability | 2 days after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative disability | 10 days after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative fatigue | Day after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative fatigue | 2 days after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative fatigue | 10 days after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative nausea | Day after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative nausea | 2 days after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative nausea | 10 days after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative complications | 10 days after surgery
  postoperative complications such as wound healing, haematoma, seroma, swelling, nausea, vomiting, bleeding, fever
Satisfaction with care | 10 days after surgery
  Satisfaction with the operation, the hospital care
Satisfaction with interventions | 10 days after surgery
  Satisfaction with the interventions

OTHER OUTCOMES:
course of surgery | day of surgery
  blood pressure, use of medication during operation, amount of gases during insufflation

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof, MD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, University of Duisburg-Essen
Locations (1):
- Abteilung für Allgemein-, Viszeral-, Gefäßchirurgie und Koloproktologie, Johanniter-Krankenhaus Rheinhausen, Duisburg, Germany

REFERENCES:
- [Background] Omlor G, Kiewitz S, Pietschmann S, Roesler S. [Effect of preoperative preoperative visualization therapy on postoperative outcome after inguinal hernia surgery and thyroid resection]. Zentralbl Chir. 2000;125(4):380-5; discussion 385-6. German. PMID 10829320